CLINICAL TRIAL: NCT04579497
Title: Temperature-dependent Changes in Cardiovascular Parameters During Warm Water Footbaths in Healthy Female Volunteers - a Blinded, Randomized, Controlled, Four-arm Study With Cross-over Design
Brief Title: Temperature-dependent Changes in Cardiovascular Parameters During Warm Water Footbaths in Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Collaborators: Universität Tübingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SWI_16
Record Dates: First submitted 2020-09-29; First posted 2020-10-08 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Warm Footbath; Cardiovascular System; Autonomic Nervous System
Keywords: Warm water footbath; Temperature-dependent effects; Cardiovascular System; Autonomic Nervous System; Heart Rate Variability; Healthy female volunteers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 38° C footbath (Experimental): Footbath with warm water at a constant temperature of 38° C
  Interventions: Other: 38°C warm water footbath
- 40° C footbath (Experimental): Footbath with warm water at a constant temperature of 40° C
  Interventions: Other: 40°C warm water footbath
- 42° C footbath (Experimental): Footbath with warm water at a constant temperature of 42° C
  Interventions: Other: 42°C warm water footbath
- Rising temperature footbath (Experimental): Footbath with warm water rising from 38° C to 42° C
  Interventions: Other: 38-42°C rising temperature footbath

INTERVENTIONS:
Other: 38°C warm water footbath — A ten-minute pre-intervention rest period followed by a 30-minute footbath with 16 l of warm water at a constant temperature of 38°C, followed by a ten-minute post-intervention rest period.
  Arms: 38° C footbath
Other: 40°C warm water footbath — A ten-minute pre-intervention rest period followed by a 30-minute footbath with 16 l of warm water at a constant temperature of 40°C, followed by a ten-minute post-intervention rest period.
  Arms: 40° C footbath
Other: 42°C warm water footbath — A ten-minute pre-intervention rest period followed by a 30-minute footbath with 16 l of warm water at a constant temperature of 42°C, followed by a ten-minute post-intervention rest period.
  Arms: 42° C footbath
Other: 38-42°C rising temperature footbath — A ten-minute pre-intervention rest period followed by a 30-minute footbath with 16 l of warm water. Water temperature starts at 38°C and is increased by 1°C every 6 minutes, resulting in 42°C after 30 minutes. The footbath is followed by a ten-minute post-intervention rest period.
  Arms: Rising temperature footbath

SUMMARY:
A study to explore whether different temperatures of warm water footbaths have different effects on the cardiovascular system, the autonomic nervous system and the general well-being of healthy women.

DETAILED DESCRIPTION:
This is a blinded, four-arm randomized controlled trial with crossover design to explore the effects of warm water footbaths with different water temperatures on cardiovascular stress, reaction of the autonomic nervous system and a feeling of comfort and warmth in healthy female volunteers. Cardiovascular and ANS measurements are performed continuously throughout the interventions and the participants rate their feelings of warmth, general well-being and the footbath-related comfort with questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age between 18 and 55 years

Exclusion Criteria:

* Male sex
* Chronic skin lesions at the lower legs or feet
* Varicose veins grade 3 and grade 4 (Marshall stage classification), chronic venous insufficiency
* Cardiac arrhythmia
* Cardiac pacemaker
* Asthma bronchiale
* Consumption of HRV-modulating medication (especially tricyclic antidepressants, beta blockers)
* Pregnancy
* Insufficient knowledge of the German language

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Pressure Rate Product (PRP) at timepoint t5 (footbath minute 21-30) | Timepoint 5 (t5 = mean of the measurements recorded from minute 21-30 of the 30-minute footbath)
  Pressure Rate Product (PRP), calculated from systolic blood pressure (measured with the Mobil-O-Graph® PWA) and heart rate (measured with the Bittium Faros 360TM ECG recorder) at timepoint 5 (t5 = mean of the measurements recorded from minute 21 to minute 30 of the footbath).

SECONDARY OUTCOMES:
Change in Pressure Rate Product (PRP) at timepoints t1 (minute 1-10 of the pre-intervention rest period), t3 (minute 1-10 of the footbath), t4 (minute 11-20 of the footbath), and t7 (minute 1-10 of the post-intervention rest period). | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Pressure Rate Product (PRP), calculated from systolic blood pressure (measured with the Mobil-O-Graph® PWA) and heart rate (measured with the Bittium Faros 360TM ECG recorder) at timepoints t1 (t1 = mean of the measurements recorded from minute 1 to minute 10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1 to minute 10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11 to minute 20 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1 to minute 10 of the post-intervention rest period).
Heart rate variability (HRV) analysis: Change in SDNN | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  SDNN: Standard deviation of normal to normal (NN) intervals (ms) (Bittium Faros 360TM ECG recorder). Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in pNN50 | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  pNN50: Percentage of successive NN intervals that differ from each other by more than 50 ms (%) (Bittium Faros 360TM ECG recorder). Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in HF | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  HF: High frequency power band (0.15-0.40 Hz) (ms2) from frequency domain analysis (Bittium Faros 360TM ECG recorder). Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in LF | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  LF: Low frequency power band (0.04-0.15 Hz) (ms2) from frequency domain analysis (Bittium Faros 360TM ECG recorder). Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in LF/HF ratio | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  LF/HF ratio = ratio of two bands from frequency domain analysis: LF band (0.04-0.15 Hz), HF band (0.15-0.40 Hz) (Bittium Faros 360TM ECG recorder). Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in VLF | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  VLF: Very low frequency power band (0.0033-0.04 Hz) (ms2) from frequency domain analysis (Bittium Faros 360TM ECG recorder). Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Mean Heart Rate | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Mean heart rate (bpm) (Bittium Faros 360TM ECG recorder). Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in SD2/SD1 ratio | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  SD2/SD1 ratio, derived from Poincaré plot (Bittium Faros 360TM ECG recorder). Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Stress Index | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Stress Index (SI) according to Baevsky's formula SI = AMo/2Mo*MxDMn (Mo = mode, AMo = mode amplitude, MxDMn = variation range of RR intervals) (Bittium Faros 360TM ECG recorder). Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Respiration Rate | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Respiration rate (1/min) (Bittium Faros 360TM ECG recorder). Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Heart Rate/Respiration Rate ratio | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Heart rate/respiration rate ratio (Bittium Faros 360TM ECG recorder). Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in RMSSD | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  RMSSD: Root mean square of successive differences (ms) (Bittium Faros 360TM ECG recorder). Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Stiffness Index | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Stiffness Index, measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Perfusion Index | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Perfusion Index, measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Peak to Peak Time | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Peak to Peak Time (PPT, ms), measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in SlopeInW1 | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  SlopeInW1, measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in SlopeInW2 | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  SlopeInW2, measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in SlopeInW3 | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  SlopeInW3, measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in SlopeInW4 | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  SlopeInW4, measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Reflection Index | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Reflection Index, measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in TimeTX | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  TimeTX (ms), measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in TimeTY | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  TimeTY (ms), measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in QuotTYTX | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  QuotTYTX, measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in AreaAX | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  AreaAX, measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in AreaAY | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  AreaAY, measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in QuotAYAX | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  QuotAYAX, measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in TimeTV | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  TimeTV (ms), measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in TimeTW | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  TimeTW (ms), measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in QuotTVTW | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  QuotTVTW, measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in AreaAV | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  AreaAV, measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in AreaAW | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  AreaAW, measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in QuotAVAW | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  QuotAVAW, measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Oxygen Saturation | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Oxygen saturation (SpO2, %), measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Pulse Transit Time | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Pulse Transit Time (PTT, ms), measured with the Vitaguard® VG 3100 monitor, getemed, Germany. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Systolic Blood Pressure | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Systolic Blood Pressure (mmHg), measured with the Mobil-O-Graph® PWA. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Diastolic Blood Pressure | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Diastolic Blood Pressure (mmHg), measured with the Mobil-O-Graph® PWA. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Mean Arterial Pressure | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Mean Arterial Pressure (mmHg), measured with the Mobil-O-Graph® PWA. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Pulse Pressure | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Pulse Pressure (mmHg), measured with the Mobil-O-Graph® PWA. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Stroke Volume | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Stroke Volume (ml), measured with the Mobil-O-Graph® PWA. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Cardiac Output | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Cardiac Output (l/min), measured with the Mobil-O-Graph® PWA. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Peripheral Resistance | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Peripheral Resistance, measured with the Mobil-O-Graph® PWA. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Cardiac Index | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Cardiac Index, measured with the Mobil-O-Graph® PWA. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Augmentation Pressure | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Augmentation Pressure (mmHg), measured with the Mobil-O-Graph® PWA. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Augmentation Index | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Augmentation Index, measured with the Mobil-O-Graph® PWA. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in Pulse Wave Velocity | Physiological parameters are measured continuously (Vitaguard® VG 3100, GETEMED; Bittium Faros 360TM) and every 2 min (Mobil-O-Graph® PWA) for a total duration of 50 min.
  Pulse Wave Velocity (PWV, m/s), measured with the Mobil-O-Graph® PWA. Measurements analysed at timepoints t1 (t1 = mean of the measurements recorded from minute 1-10 of the pre-intervention rest period), t3 (t3 = mean of the measurements recorded from minute 1-10 of the footbath), t4 (t4 = mean of the measurements recorded from minute 11-20 of the footbath), t5 (t5 = mean of the measurements recorded from minute 21-30 of the footbath), and t7 (t7 = mean of the measurements recorded from minute 1-10 of the post-intervention rest period).
Change in warmth perception at the feet | Immediately before (timepoint 2, t2), immediately after (timepoint 6, t6) and 10 minutes following the footbath (timepoint 8, t8) (length of footbath is up to 30 minutes).
  Self-reported warmth perception at both feet, assessed with the "Herdecke warmth perception questionnaire" immediately before (timepoint 2, t2), immediately after (timepoint 6, t6) and 10 minutes following the footbath (timepoint 8, t8). Each item is scored 0-4 (0 = cold; 4 = hot), yielding a mean between 0 and 4.
Change in warmth perception at the hands | Immediately before (timepoint 2, t2), immediately after (timepoint 6, t6) and 10 minutes following the footbath (timepoint 8, t8) (length of footbath is up to 30 minutes).
  Self-reported warmth perception at both hands, assessed with the "Herdecke warmth perception questionnaire" immediately before (timepoint 2, t2), immediately after (timepoint 6, t6) and 10 minutes following the footbath (timepoint 8, t8). Each item is scored 0-4 (0 = cold; 4 = hot), yielding a mean between 0 and 4.
Change in warmth perception at the head | Immediately before (timepoint 2, t2), immediately after (timepoint 6, t6) and 10 minutes following the footbath (timepoint 8, t8) (length of footbath is up to 30 minutes).
  Self-reported warmth perception at the head, assessed with the "Herdecke warmth perception questionnaire" immediately before (timepoint 2, t2), immediately after (timepoint 6, t6) and 10 minutes following the footbath (timepoint 8, t8). Each item is scored 0-4 (0 = cold; 4 = hot), yielding a mean between 0 and 4.
Change in overall warmth perception | Immediately before (timepoint 2, t2), immediately after (timepoint 6, t6) and 10 minutes following the footbath (timepoint 8, t8) (length of footbath is up to 30 minutes).
  Self-reported overall warmth perception, assessed with the "Herdecke warmth perception questionnaire" immediately before (timepoint 2, t2), immediately after (timepoint 6, t6) and 10 minutes following the footbath (timepoint 8, t8). The item is scored 0-4 (0 = cold; 4 = hot).
Change in general well-being | Immediately before (timepoint 2, t2), immediately after (timepoint 6, t6) and 10 minutes following the footbath (timepoint 8, t8) (length of footbath is up to 30 minutes).
  Self-reported well-being, assessed with the "Basler Befindlichkeits-Skala" (Basel Mood Questionnaire, BBS) immediately before (t2), immediately after (t6) and 10 minutes following the footbath (t8) (BBS: 16 items; 7-point rating scale; higher values represent a better outcome).
Change in feeling of comfort during footbath | Immediately before the footbath (timepoint 2, t2), every 6 minutes during the 30-minute footbath, and 10 minutes following the footbath (timepoint 8, t8).
  Self-reported footbath comfort, assessed with a 7-point face scale ranging from "very comfortable" (laughing face) to "very hard stress" (crying face).

OTHER OUTCOMES:
Change in warmth perception and skin stimulus at the feet during the footbath | Up to 30 minutes.
  Self-reported perception of warmth and skin stimulus during the footbath, assessed with a dynamic warmth and skin stimulus visual analog scale (VAS), applied once per minute (0 = cold/no stimulus; 10 = very hot/very strong stimulus).
Preferred footbath | 10 minutes.
  Self-reported personal preference of footbath, assessed with a short questionnaire asking which footbath had the most positive overall effect (check boxes to mark for the first, second, third, or fourth footbath) and why (short, self-formulated statement of reasons). Assessed once after the fourth footbath intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, Dr, Principal Investigator — Arcim Institute
Locations (1):
- Arcim Institute, Filderstadt, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available, in addition to study protocol and informed consent form.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available upon publication for a duration of three months.
Access Criteria: The data will be made available to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.